CLINICAL TRIAL: NCT05372081
Title: Clinical and Molecular Study With Digital Support of Patients With Inoperable Lung Cancer
Acronym: SNF-CLIMEDIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Stavros Niarchos Foundation (Unknown); Care Across Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: HE2SN/21
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Non-Small Cell Carcinoma of Lung, TNM Stage 4
Keywords: observational study; digital platform
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and Formalin Fixed Paraffin Embedded tumour tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who will receive digital assistant: Patients will receive digital assistance (in a few words text format) for any symptoms/adverse events they will include in their profile in the digital platform.
  Interventions: Other: Digital platform
- Patients who will not receive digital assistant: Patients will just include any symptoms/adverse events in their profile in the digital platform.
  Interventions: Other: Digital platform

INTERVENTIONS:
Other: Digital platform — Patients will be randomized (1:1) in the way they will receive or not any assistance from the digital platform.

SUMMARY:
The purpose of this study is to provide high quality oncology services to patients with inoperable Non-Small Cell Lung Cancer (NSCLC) in Greece. These services will be based on 3 pillars:

1. Clinical: personalized treatment will be administered and its effectiveness and safety will be recorded and evaluated.
2. Molecular: the gene footprint of each patient at the beginning of his treatment, the molecular identity of his tumor will be analyzed and recorded based on analysis with modern Next Generation Sequencing (NGS) techniques.
3. Digital: Patients will have access to the digital platform where they will record the adverse reactions they will face during their treatment.

DETAILED DESCRIPTION:
Lung cancer is the primary cause of cancer death worldwide regardless of gender or age group. Based on the most recent statistics for our country, every year about 9000 new cases of lung cancer are diagnosed. Lung cancer is the most common type of cancer in Greece in both men and women. It is estimated that about 8000 people lose their lives annually from this disease, while the total number of deaths from lung cancer seems to exceed in number the sum of deaths due to breast, prostate and colorectal cancer.

For many decades chemotherapy was the cornerstone and the only treatment option for lung cancer. In the last 20 years, the discovery and study of various molecular subtypes in non-small cell lung cancer has led to the development of targeted therapies. Modern oncology has multiple targeted therapies for corresponding molecular subtypes, such as ROS-1 rearrangements, amplifications and mutations of the MET gene, RET rearrangements, mutations of the BRAF gene, NTRK gene fusions, HER2 gene mutations, as well as KRAS mutations.The detection of molecular pathways, targeted mutations and biomarkers is a critical step in the diagnosis and treatment of patients with non-small cell lung cancer, in both early and advanced stage.The use of NGS (Next Generation Sequencing) technology as modern tool for accessing genetic material is adopted by more and more clinicians worldwide. The molecular analysis of the tumor with the technique of NGS, is considered as a necessity in the practice of modern oncology in order the patients to receive the best treatments for their disease.

a) Clinical pillar: In this study will be included 200 patients, 18 years old and older, with PS 0-2, treated for inoperable NSCLC stage IV. Patient will be treated according to the local standard of care based on their medical history. b)After signing the Informed Consent patients will provide biological material (blood samples and Formalin fixed paraffin embedded tissues) in order to proceed with the molecular arm of the study and the extended NGS analysis. In addition to molecular analysis, an economic analysis of the use of health resources will follow for a detailed understanding of the relevant financial aggregates and the improvement of the performance of existing resources. c) On the digital arm each patient will have access in the digital platform of CAREACCROSS which allows continuous and remote access for both patient and their physician with absolute security and data privacy.

All patients will be included in the digital monitoring and information program from their mobile phone and will have contact the investigator and the study team.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-small cell lung cancer stage IV
* No younger than 18 years old patients
* Performance status: 0-2
* Existence of biological material for the molecular analysis
* Patients who have not been treated with any other treatment than adjuvant
* Ability to use a mobile device or computer for digital communication

Exclusion Criteria:

* Childbearing women
* Patients with PS > 3
* Limited ability to use a mobile device for basic digital communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non- Small Cell Lung Cancer candidates for 1st- line treatment (or previously having received adjuvant therapy), available FFPE tissue and blood sample and able to use a mobile device for basic digital communication
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Molecular identification of patients with non-small cell lung cancer | up to 36 months

SECONDARY OUTCOMES:
Overall survival | up to 36 months
Data correlation | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Paris Kosmidis, MD, Principal Investigator — YGEIA Hospital
Locations (15):
- Greece (15):
  - Ygeia Hospital, Psychikó, Attica
  - MITERA Hospital, Athens, Marousi
  - General University Hospital of Larissa, Larissa, Mezourlo
  - 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens, Nea Kifisia
  - 4th Dept of Medical Oncology, Metropolitan Hospital, Athens, Neo Faliro
  - Henry Dunant Hospital Center, Athens
  - EUROCLINIC of Athens, Athens
  - 401 General Military Hospital of Athens, Athens
  - 1st Dept of Medical Oncology, Metropolitan Hospital, Athens
  - 2nd Dept of Medical Oncology, Metropolitan Hospital, Athens
  - General Hospital of Kavalas, Kavala
  - General Hospital of Patra "Agios Andreas", Pátrai
  - Division of Oncology, Dept of Internal Medicine, University Hospital of Patras, Pátrai
  - 2nd Dept of Medical Oncology, EUROMEDICA General Clinic of Thessaloniki, Thessaloniki
  - General Hospital of Thessalonikis "G. Papanikolaou", Thessaloniki

REFERENCES:
- [Background] Fountzilas G, Giannoulatou E, Alexopoulou Z, Zagouri F, Timotheadou E, Papadopoulou K, Lakis S, Bobos M, Poulios C, Sotiropoulou M, Lyberopoulou A, Gogas H, Pentheroudakis G, Pectasides D, Koutras A, Christodoulou C, Papandreou C, Samantas E, Papakostas P, Kosmidis P, Bafaloukos D, Karanikiotis C, Dimopoulos MA, Kotoula V. TP53 mutations and protein immunopositivity may predict for poor outcome but also for trastuzumab benefit in patients with early breast cancer treated in the adjuvant setting. Oncotarget. 2016 May 31;7(22):32731-53. doi: 10.18632/oncotarget.9022. PMID 27129168
- [Background] Rothberg JM, Hinz W, Rearick TM, Schultz J, Mileski W, Davey M, Leamon JH, Johnson K, Milgrew MJ, Edwards M, Hoon J, Simons JF, Marran D, Myers JW, Davidson JF, Branting A, Nobile JR, Puc BP, Light D, Clark TA, Huber M, Branciforte JT, Stoner IB, Cawley SE, Lyons M, Fu Y, Homer N, Sedova M, Miao X, Reed B, Sabina J, Feierstein E, Schorn M, Alanjary M, Dimalanta E, Dressman D, Kasinskas R, Sokolsky T, Fidanza JA, Namsaraev E, McKernan KJ, Williams A, Roth GT, Bustillo J. An integrated semiconductor device enabling non-optical genome sequencing. Nature. 2011 Jul 20;475(7356):348-52. doi: 10.1038/nature10242. PMID 21776081
- [Background] Hovelson DH, McDaniel AS, Cani AK, Johnson B, Rhodes K, Williams PD, Bandla S, Bien G, Choppa P, Hyland F, Gottimukkala R, Liu G, Manivannan M, Schageman J, Ballesteros-Villagrana E, Grasso CS, Quist MJ, Yadati V, Amin A, Siddiqui J, Betz BL, Knudsen KE, Cooney KA, Feng FY, Roh MH, Nelson PS, Liu CJ, Beer DG, Wyngaard P, Chinnaiyan AM, Sadis S, Rhodes DR, Tomlins SA. Development and validation of a scalable next-generation sequencing system for assessing relevant somatic variants in solid tumors. Neoplasia. 2015 Apr;17(4):385-99. doi: 10.1016/j.neo.2015.03.004. PMID 25925381
- [Background] Luthra R, Patel KP, Routbort MJ, Broaddus RR, Yau J, Simien C, Chen W, Hatfield DZ, Medeiros LJ, Singh RR. A Targeted High-Throughput Next-Generation Sequencing Panel for Clinical Screening of Mutations, Gene Amplifications, and Fusions in Solid Tumors. J Mol Diagn. 2017 Mar;19(2):255-264. doi: 10.1016/j.jmoldx.2016.09.011. Epub 2016 Dec 23. PMID 28017569
- [Background] Mehrotra M, Duose DY, Singh RR, Barkoh BA, Manekia J, Harmon MA, Patel KP, Routbort MJ, Medeiros LJ, Wistuba II, Luthra R. Versatile ion S5XL sequencer for targeted next generation sequencing of solid tumors in a clinical laboratory. PLoS One. 2017 Aug 2;12(8):e0181968. doi: 10.1371/journal.pone.0181968. eCollection 2017. PMID 28767674
- [Background] Dehghani M, Rosenblatt KP, Li L, Rakhade M, Amato RJ. Validation and Clinical Applications of a Comprehensive Next Generation Sequencing System for Molecular Characterization of Solid Cancer Tissues. Front Mol Biosci. 2019 Sep 25;6:82. doi: 10.3389/fmolb.2019.00082. eCollection 2019. PMID 31681791
- [Background] Lih CJ, Harrington RD, Sims DJ, Harper KN, Bouk CH, Datta V, Yau J, Singh RR, Routbort MJ, Luthra R, Patel KP, Mantha GS, Krishnamurthy S, Ronski K, Walther Z, Finberg KE, Canosa S, Robinson H, Raymond A, Le LP, McShane LM, Polley EC, Conley BA, Doroshow JH, Iafrate AJ, Sklar JL, Hamilton SR, Williams PM. Analytical Validation of the Next-Generation Sequencing Assay for a Nationwide Signal-Finding Clinical Trial: Molecular Analysis for Therapy Choice Clinical Trial. J Mol Diagn. 2017 Mar;19(2):313-327. doi: 10.1016/j.jmoldx.2016.10.007. Epub 2017 Feb 7. PMID 28188106
- [Background] El-Deiry WS, Goldberg RM, Lenz HJ, Shields AF, Gibney GT, Tan AR, Brown J, Eisenberg B, Heath EI, Phuphanich S, Kim E, Brenner AJ, Marshall JL. The current state of molecular testing in the treatment of patients with solid tumors, 2019. CA Cancer J Clin. 2019 Jul;69(4):305-343. doi: 10.3322/caac.21560. Epub 2019 May 22. PMID 31116423
- [Background] Duma N, Santana-Davila R, Molina JR. Non-Small Cell Lung Cancer: Epidemiology, Screening, Diagnosis, and Treatment. Mayo Clin Proc. 2019 Aug;94(8):1623-1640. doi: 10.1016/j.mayocp.2019.01.013. PMID 31378236
- [Background] Friedlaender A, Bauml J, Banna GL, Addeo A. Identifying successful biomarkers for patients with non-small-cell lung cancer. Lung Cancer Manag. 2019 Nov 14;8(3):LMT17. doi: 10.2217/lmt-2019-0009. No abstract available. PMID 31807145
- [Background] Osei, E., Lumini, J., Gunasekara, D., Osei, B., Asare, A., & Laflamme, R. (2020). A review of predictive, prognostic and diagnostic biomarkers for non-small-cell lung cancer: Towards personalised and targeted cancer therapy. Journal of Radiotherapy in Practice, 19(4), 370-384. doi:10.1017/S1460396919000876
- [Background] Heeke AL, Pishvaian MJ, Lynce F, Xiu J, Brody JR, Chen WJ, Baker TM, Marshall JL, Isaacs C. Prevalence of Homologous Recombination-Related Gene Mutations Across Multiple Cancer Types. JCO Precis Oncol. 2018;2018:PO.17.00286. doi: 10.1200/PO.17.00286. Epub 2018 Jul 23. PMID 30234181
- [Background] Kandoth C, McLellan MD, Vandin F, Ye K, Niu B, Lu C, Xie M, Zhang Q, McMichael JF, Wyczalkowski MA, Leiserson MDM, Miller CA, Welch JS, Walter MJ, Wendl MC, Ley TJ, Wilson RK, Raphael BJ, Ding L. Mutational landscape and significance across 12 major cancer types. Nature. 2013 Oct 17;502(7471):333-339. doi: 10.1038/nature12634. PMID 24132290
- [Background] Knijnenburg TA, Wang L, Zimmermann MT, Chambwe N, Gao GF, Cherniack AD, Fan H, Shen H, Way GP, Greene CS, Liu Y, Akbani R, Feng B, Donehower LA, Miller C, Shen Y, Karimi M, Chen H, Kim P, Jia P, Shinbrot E, Zhang S, Liu J, Hu H, Bailey MH, Yau C, Wolf D, Zhao Z, Weinstein JN, Li L, Ding L, Mills GB, Laird PW, Wheeler DA, Shmulevich I; Cancer Genome Atlas Research Network; Monnat RJ Jr, Xiao Y, Wang C. Genomic and Molecular Landscape of DNA Damage Repair Deficiency across The Cancer Genome Atlas. Cell Rep. 2018 Apr 3;23(1):239-254.e6. doi: 10.1016/j.celrep.2018.03.076. PMID 29617664
- [Background] Ricciuti B, Recondo G, Spurr LF, Li YY, Lamberti G, Venkatraman D, Umeton R, Cherniack AD, Nishino M, Sholl LM, Shapiro GI, Awad MM, Cheng ML. Impact of DNA Damage Response and Repair (DDR) Gene Mutations on Efficacy of PD-(L)1 Immune Checkpoint Inhibition in Non-Small Cell Lung Cancer. Clin Cancer Res. 2020 Aug 1;26(15):4135-4142. doi: 10.1158/1078-0432.CCR-19-3529. Epub 2020 Apr 24. PMID 32332016
- [Background] Pfarr N, Kirchner M, Lehmann U, Leichsenring J, Merkelbach-Bruse S, Glade J, Hummel M, Stogbauer F, Lehmann A, Trautmann M, Kumbrink J, Jung A, Dietmaier W, Endris V, Kazdal D, Evert M, Horst D, Kreipe H, Kirchner T, Wardelmann E, Lassen U, Buttner R, Weichert W, Dietel M, Schirmacher P, Stenzinger A. Testing NTRK testing: Wet-lab and in silico comparison of RNA-based targeted sequencing assays. Genes Chromosomes Cancer. 2020 Mar;59(3):178-188. doi: 10.1002/gcc.22819. Epub 2019 Nov 18. PMID 31652375